CLINICAL TRIAL: NCT05372224
Title: Vitamin D Improves Osteoporosis in Postmenopausal Women With Denosumab Failure
Brief Title: Effect of Vitamin D and Denosumab on Bone Remodelling in Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Regional 1o de Octubre (Other)
Collaborators: Universidad Nacional Autonoma de Mexico (Other); National Polytechnic Institute, Mexico (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 032.2020
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Hypovitaminosis D; Osteoporosis, Postmenopausal; Menopause
Keywords: Vitamin D; Postmenopausal Osteoporosis; Denosumab; Hypovitaminosis D; Osteoporosis; Osteopenia
MeSH Terms: conditions — Vitamin D Deficiency; Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: 76 participants were considered from the climacteric clinic of the regional hospital "1o de Octubre" of the Institute of Security and Social Services for State Workers (ISSSTE), of which 23 presented elimination criteria, and 55 were included in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitamin D 4000 IU (Experimental): 4000 IU of vitamin D were administrated once a day orally and calcium carbonate 1.2 g a day in a single dose.
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 4000 IU were administrated once a day for 3 months.
  Other Names: Histofil®

SUMMARY:
Denosumab is a monoclonal antibody against RANKL ligand, which is used as an alternative treatment for osteoporosis in patients who have a poor response to first-line antiresorptive therapy. However, discontinuation of denosumab produces a rapid increase in bone turnover, bone loss and potentially increased risk of multiple vertebral fractures.

DETAILED DESCRIPTION:
76 postmenopausal women from the climacteric clinic of the regional hospital "1o de Octubre" of the Institute of Security and Social Services for State Workers (ISSSTE) were firstly considered, of which 23 presented elimination criteria and only 55 who had received denosumab therapy for an average of 2.5 years without a significant improvement in hip and lumbar spine T-scores were enrolled. First, a general medical evaluation was performed. Serum levels of vitamin D were analysed to find the prevalence of hypovitaminosis D. A bone mineral density test was done to calculate hip and lumbar spine T-scores. Then, vitamin D was administrated daily for one year at a dose of 4,000 IU and the studies were repeated after one year. Statistical analysis was performed using PAST 3.0 and GraphPad Prism 8.4.3. software. The arithmetic median (µ) and standard deviation (S.D.) were calculated using Excel-Word. Graphics were constructed with GraphPad Prism 8.4.3 and tables with Excel Word. Categorical variables were analysed with chi-squared or Fisher exact test depending on the number of participants in each cell. Normality was determined using the Shapiro-Wilk test. To compare two paired samples, the Wilcoxon signed-rank test was utilized. The assigned α value for this study was <0.05. In all cases, if a Montecarlo permutation was available, the exact p-value was taken instead of the raw p-value.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postmenopausal osteoporosis or osteopenia in treatment with denosumab 60mg every six months plus calcium carbonate 1.2g/day + vitamin D 800IU/day.
* Diagnosis of hypovitaminosis D, with serum cholecalciferol values <30ng/dL.

Exclusion Criteria:

* Incomplete clinical records or clinical records.
* Age over 90 years.
* Diagnosis of secondary (hereditary) osteoporosis.
* History of prolonged use of steroids.
* Lack of adherence to medical treatment.
* Diagnosis of cancer.
* Diagnosis of depression.
* Diagnosis of Celiac disease or with the presence of alterations in intestinal absorption.
* Allergies to any of the medications administered.

Ages: 45 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2021-06-22 (Actual); Study Completion 2021-06-22 (Actual)

PRIMARY OUTCOMES:
Number of participants with hip T-score improvement at 12 months | 12 months
  It refers to the number of participants who improved their hip T-score at three months after treatment.
Number of participants with lumbar spine T-score improvement at 12 months | 12 months
  It refers to the number of participants who improved their lumbar spine T-score at three months after treatment.
Number of participants with osteoporosis of the hip at 12 months | 12 months
  It refers to the number of participants that present a hip T-score above -2.5 three months after treatment.
Number of participants with osteoporosis of the lumbar spine at 12 months | 12 months
  It refers to the number of participants that present a lumbar spine T-score greater than -2.5 three months after treatment.
Number of participants with osteopenia on the hip at 12 months | 12 months
  It refers to the number of participants that present a hip T-score from -1 to -2.4 three months after treatment.
Number of participants with osteopenia of the lumbar spine at 12 months | 12 months
  It refers to the number of participants that present a lumbar spine T-score from -1 to -2.4 three months after treatment.
Number of participants with normal hip T-score at 12 months | 12 months
  It refers to the number of participants that present a hip T-score below -1 three months after treatment.
Number of participants with normal lumbar spine T-score at 12 months | 12 months
  It refers to the number of participants that present a lumbar spine T-score below -1 three months after treatment.
Number of participants with improvement in serum levels of vitamin D at 12 months | 12 months
  Improvement in serum levels of 25-hydroxy vitamin D [25(OH)D] was considered when serum vitamin D levels increased concerning baseline levels.
Number of participants with clinical remission of hypovitaminosis D at 12 months | 12 months
  Remission of hypovitaminosis D was considered when serum levels of 25-hydroxy vitamin D [25(OH)D] were above 29 pg/ml.

SECONDARY OUTCOMES:
Number of participants with vitamin D sufficiency at 12 months | 12 months
  It refers to the number of participants who reached serum levels of vitamin D above 29 pg/ml after three months of treatment.
Number of participants with vitamin D insufficiency at 12 months | 12 months
  It refers to the number of participants who reached serum levels of vitamin D of 21 to 29 pg/ml after three months of treatment.
Number of participants with vitamin D deficiency at 12 months | 12 months
  It refers to the number of participants who reached serum levels of vitamin D less than 20 pg/ml after three months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: María B Brito-Gavilanes, M.D., Principal Investigator — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1 ISSSTE; Patricia Loranca-Moreno, M.D., M.Sc., Principal Investigator — Peri-postmenopause and bone metabolism clinic. Regional Hospital October 1st ISSSTE.; Juan M Ocampo-Godínez, M.D., P.hD, Principal Investigator — Laboratory of Tissue Engineering, UNAM
Locations (1):
- Patricia Loranca-Moreno, Mexico City, Gustavo A. Madero, Mexico

REFERENCES:
- [Background] Tsourdi E, Langdahl B, Cohen-Solal M, Aubry-Rozier B, Eriksen EF, Guanabens N, Obermayer-Pietsch B, Ralston SH, Eastell R, Zillikens MC. Discontinuation of Denosumab therapy for osteoporosis: A systematic review and position statement by ECTS. Bone. 2017 Dec;105:11-17. doi: 10.1016/j.bone.2017.08.003. Epub 2017 Aug 5. PMID 28789921
- [Background] McClung MR, Wagman RB, Miller PD, Wang A, Lewiecki EM. Observations following discontinuation of long-term denosumab therapy. Osteoporos Int. 2017 May;28(5):1723-1732. doi: 10.1007/s00198-017-3919-1. Epub 2017 Jan 31. PMID 28144701
- [Background] Kanis JA, Cooper C, Rizzoli R, Reginster JY; Scientific Advisory Board of the European Society for Clinical and Economic Aspects of Osteoporosis (ESCEO) and the Committees of Scientific Advisors and National Societies of the International Osteoporosis Foundation (IOF). European guidance for the diagnosis and management of osteoporosis in postmenopausal women. Osteoporos Int. 2019 Jan;30(1):3-44. doi: 10.1007/s00198-018-4704-5. Epub 2018 Oct 15. PMID 30324412
- [Background] Miyoshi A, Kameda H, Nagai S, Nakamura A, Miya A, Takase T, Atsumi T, Miyoshi H. Beneficial effects of switching to denosumab from bisphosphonates or selective estrogen receptor modulators in postmenopausal women with type 2 diabetes and osteopenia/osteoporosis. J Diabetes Investig. 2021 Jul;12(7):1293-1300. doi: 10.1111/jdi.13458. Epub 2020 Dec 13. PMID 33141482
- [Background] Saag KG, Petersen J, Brandi ML, Karaplis AC, Lorentzon M, Thomas T, Maddox J, Fan M, Meisner PD, Grauer A. Romosozumab or Alendronate for Fracture Prevention in Women with Osteoporosis. N Engl J Med. 2017 Oct 12;377(15):1417-1427. doi: 10.1056/NEJMoa1708322. Epub 2017 Sep 11. PMID 28892457
- [Background] Cummings SR, San Martin J, McClung MR, Siris ES, Eastell R, Reid IR, Delmas P, Zoog HB, Austin M, Wang A, Kutilek S, Adami S, Zanchetta J, Libanati C, Siddhanti S, Christiansen C; FREEDOM Trial. Denosumab for prevention of fractures in postmenopausal women with osteoporosis. N Engl J Med. 2009 Aug 20;361(8):756-65. doi: 10.1056/NEJMoa0809493. Epub 2009 Aug 11. PMID 19671655
- [Background] Takeuchi T, Tanaka Y, Soen S, Yamanaka H, Yoneda T, Tanaka S, Nitta T, Okubo N, Genant HK, van der Heijde D. Effects of the anti-RANKL antibody denosumab on joint structural damage in patients with rheumatoid arthritis treated with conventional synthetic disease-modifying antirheumatic drugs (DESIRABLE study): a randomised, double-blind, placebo-controlled phase 3 trial. Ann Rheum Dis. 2019 Jul;78(7):899-907. doi: 10.1136/annrheumdis-2018-214827. Epub 2019 Apr 29. PMID 31036625